CLINICAL TRIAL: NCT05025917
Title: Assessing the Effect of Shatavari Supplementation on Bone and Skeletal Muscle Health in Healthy Postmenopausal Women: A Randomised Double Blind Clinical Trial
Brief Title: Assessing the Effect of Shatavari Supplementation on Bone and Skeletal Muscle Health in Healthy Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Principal Investigator, Mary O'Leary, Research Fellow, University of Exeter
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 190206/B/01
Record Dates: First submitted 2021-08-11; First posted 2021-08-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Muscle Weakness; Osteoporosis, Postmenopausal
MeSH Terms: conditions — Muscle Weakness; Osteoporosis, Postmenopausal | interventions — stearic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shatavari (Experimental): 1000 mg per day shatavari root powder (2 x 500 mg opaque capsules; equivalent to 26,500 mg fresh weight shatavari). Ingested in the morning, daily for 6 weeks.
  Interventions: Dietary Supplement: Shatavari
- Placebo (Placebo Comparator): 1000 mg per day magnesium stearate powder (2 x 500 mg opaque capsules). Ingested in the morning, daily for 6 weeks.
  Interventions: Dietary Supplement: Magnesium stearate

INTERVENTIONS:
Dietary Supplement: Shatavari — Shatavari root powder
  Other Names: Asparagus Racemosus
  Arms: Shatavari
Dietary Supplement: Magnesium stearate — Magnesium stearate powder
  Arms: Placebo

SUMMARY:
Shatavari is a plant that grows in Nepal, Sri Lanka, India and the Himalayas and its root has long been used in Ayurvedic medicine. Its traditional uses include supporting women's health, particularly during breastfeeding and during the perimenopausal period. Shatavari has been found to contain substances that have similar chemical properties to estrogen. A decrease in the amount of ovarian estrogen production causes the menopause and this reduction in circulating estrogen has widespread effects, including promoting a decrease in bone density. This increases the risk of bone fractures. Having less oestrogen is also thought to contribute to a loss of muscle strength in postmenopausal women.

As shatavari may act on the body's tissues in a similar way to estrogen, shatavari supplementation may represent one way of preventing postmenopausal bone and muscle loss. This study will investigate these questions. 24 healthy postmenopausal women aged 60 years or older will be recruited. The participants will be randomly assigned to consume shatavari (1000 mg per day, equivalent to 26,500 mg per day fresh weight shatavari) or placebo (1000 mg per day magnesium stearate) for 6 weeks. Handgrip and knee extensor strength will be measured at baseline and at 6 weeks. Vastus lateralis (VL) muscle biopsy samples will be obtained at baseline and at 6 weeks and analysed for markers of muscle function and protein turnover. Plasma and serum samples will be collected via venepuncture and markers of bone turnover (P1NP, β-CTX) will be measured at baseline and at 6 weeks. Primary human osteoblasts (not obtained from these participants) will be stimulated with pooled sera from the placebo and shatavari supplementation conditions to assess markers of osteoblast (bone-building) activity.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (Last menstrual period > 12 months ago)
* Aged 60 years or older

Exclusion Criteria:

* BMI ≥ 30
* Diagnosis (DEXA t-score < -2.5) and/or treatment for the prevention of osteoporosis, including treatmeat with bisphosphonates and non-bisphosphonates (including, but not limited to raloxifene, denosumab, teriparatide, calcitriol and estrogenic hormone replacement therapy).
* Currently taking estrogenic hormone replacement therapy or history of estrogenic hormone replacement therapy in the past 5 years via any route of administration apart from vaginal.
* PAR-Q+ screening indicates physical activity is unsuitable.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Change in protein expression of myogenin in vastus lateralis skeletal muscle samples. | Change from baseline myogenin expression at 6 weeks.
  Measured via immunoblotting.

SECONDARY OUTCOMES:
Change in plasma concentration of markers of bone turnover. | Change from baseline concentration at 6 weeks.
  P1NP and β-CTX.
Change in plasma concentration of markers of inflammation. | Change from baseline concentration at 6 weeks.
  C-reactive protein and IL-6.
Change in handgrip strength. | Change from baseline strength at 6 weeks.
  Assessed using a handgrip dynamometer, measured in kilograms.
Change in isometric knee extensor strength | Change from baseline strength at 6 weeks.
  Assesed using an isokinetic dynamometer, measured in Newtons.
Change in isokinetc knee extensor strength | Change from baseline strength at 6 weeks.
  Assesed using an isokinetic dynamometer, measured in Newtons.

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Leary, Principal Investigator — University of Exeter
Locations (1):
- Deparment of Sport and Health Sciences, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are no plans to make IPD available. However, deidentified IPD may be made available to other researchers, on reasonable request to the Principal Investigator, provided this can be done in compliance with General Data Protection Regulations.

REFERENCES:
- [Derived] O'Leary MF, Jackman SR, Bowtell JL. Shatavari supplementation in postmenopausal women alters the skeletal muscle proteome and pathways involved in training adaptation. Eur J Nutr. 2024 Apr;63(3):869-879. doi: 10.1007/s00394-023-03310-w. Epub 2024 Jan 12. PMID 38214710